CLINICAL TRIAL: NCT01545414
Title: Internet-based CBT for Depression and Anxiety in Parkinson's Disease: a Pilot Study and Randomized Controlled Trial
Brief Title: Internet-CBT (Cognitive Behavioral Therapy) for Depression and Anxiety in Parkinsons Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICBT Parkinson
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease; Depression; Anxiety; Insomnia
Keywords: Self-help treatment; Internet treatment; Cognitive Behavioral Therapy; Internet-based Cognitive Behavioral Therapy
MeSH Terms: conditions — Parkinson Disease; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICBT (Experimental): Internet-based Cognitive Behavioral Therapy with a focus on behavioral activation
  Interventions: Behavioral: ICBT
- ICONTROL (Active Comparator): Internet-based treatment with a focus on relaxation training
  Interventions: Behavioral: ICONTROL
- SMT (No Intervention): Standard Medical Treatment while being on the waitlist for randomization to any of the active treatments

INTERVENTIONS:
Behavioral: ICBT — 12 weeks of Internet-based Cognitive Behavioral Therapy with a focus on behavioral activation
  Arms: ICBT
Behavioral: ICONTROL — 12 weeks of Internet-based treatment with a focus on relaxation training
  Arms: ICONTROL

SUMMARY:
The purpose of this project is to develop and evaluate Internet-based Cognitive Behavioral Therapy (ICBT) for Parkinson's Disease (PD) patients with concurrent depression or anxiety symptoms. All treatment in this project is given as an adjunct to Standard Medical Treatment (SMT). ICBT will be compared to an Internet-based active control treatment (ICONTROL) and to SMT alone. It is hypothesized that both active treatments will be superior to SMT, and that ICBT will be superior to ICONTROL, in reducing symptoms of depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease
* At least mild to moderate depression or anxiety defined as HADS-A or HADS-D > 7

Exclusion Criteria:

* Has a high alcohol or drug use assessed by the AUDIT / DUDIT and assessment interview
* Somatic or psychiatric problems that are directly contraindicated or seriously hamper the implementation of the treatment (eg, psychotic disorders or bipolar disorder)
* Difficulties that hamper the use of a computer
* The patient states difficulties in finding enough time for treatment
* Too low cognitive functioning defined as MoCA < 24
* Too severe depression, defined as MADRS-S over 30
* Too high suicidal risk defined as more than 4 points on the MADRS-S question 9 or according to the structured assessment interview

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in HADS | 12 weeks (Post), 3 and 6 months (FU)
  Hospital Anxiety and Depression Scale - self rating, to measure anxiety and depression

SECONDARY OUTCOMES:
Change (from baseline) in MADRS-S | 12 weeks (Post), 3 and 6 months (FU)
  Montgomery and Asberg Depressions Rating Scale - Self report, to measure level of depression
Change (from baseline) in ISI | 12 weeks (Post), 3 and 6 months (FU)
  Insomnia Severity Index - self-report, to measure insomnia symptoms
Change (from baseline) in PDQ-8 | 12 weeks (Post), 3 and 6 months (FU)
  The Parkinson's Disease Questionnaire-8, to measure various health aspects specific for PD patients
Change (from baseline) in EQ-5D | 12 weeks (Post), 3 and 6 months (FU)
  EQ-5D, to measure general health and quality of life
Change (from baseline) in SDS | 12 weeks (Post), 3 and 6 months (FU)
  Sheehan Disability Scale, to measure everyday level of functioning
Change (from baseline) in NMSQuest | 12 weeks (Post), 3 and 6 months (FU)
  Non-Motor Symptoms Questionnaire, to measure the non-motor symptoms in PD

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienehten (Internet Psychiatry Unit), Psykiatri Sydväst, SLSO, Stockholm, Sweden

REFERENCES:
- See also: The public page of the Internet-CBT treatment platform — http://www.internetpsykiatri.se